CLINICAL TRIAL: NCT05122143
Title: Pivotal, Randomized, Open-Label, 3-Period Crossover Study to Assess the Efficacy and Safety of AM-301 on Allergic Symptoms During House Dust Mite Challenge in an Exposure Chamber in Study Participants With Perennial Allergic Rhinitis
Brief Title: Efficacy and Safety of AM-301 on Allergic Symptoms of Perennial Allergic Rhinitis Sufferers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altamira Medica Ltd. (Industry)
Responsible Party: Sponsor
Organization: Auris Medical, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AM-301-CL-21-02
Record Dates: First submitted 2021-10-26; First posted 2021-11-16 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Perennial Allergic Rhinitis; Rhinitis, Allergic
Keywords: Allergic rhinitis symptoms; Runny nose; Itchy nose
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic; Rhinorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Treatment sequence for the 3 treatment exposure visits is ABC.
  Interventions: Device: Treatment A; Device: Treatment B; Other: Treatment C
- Sequence 2 (Experimental): Treatment sequence for the 3 treatment exposure visits is BCA.
  Interventions: Device: Treatment A; Device: Treatment B; Other: Treatment C
- Sequence 3 (Experimental): Treatment sequence for the 3 treatment exposure visits is CAB.
  Interventions: Device: Treatment A; Device: Treatment B; Other: Treatment C
- Sequence 4 (Experimental): Treatment sequence for the 3 treatment exposure visits is ACB.
  Interventions: Device: Treatment A; Device: Treatment B; Other: Treatment C
- Sequence 5 (Experimental): Treatment sequence for the 3 treatment exposure visits is BAC.
  Interventions: Device: Treatment A; Device: Treatment B; Other: Treatment C
- Sequence 6 (Experimental): Treatment sequence for the 3 treatment exposure visits is CBA.
  Interventions: Device: Treatment A; Device: Treatment B; Other: Treatment C

INTERVENTIONS:
Device: Treatment A — Nasal Spray with drug-free aqueous gel emulsion (AM-301) intended to help protect against airborne allergens.
  One Spray of AM-301 per nostril
  Other Names: Bentrio
Device: Treatment B — Nasal Spray with drug-free aqueous gel emulsion (AM-301) intended to help protect against airborne allergens.
  Two Sprays of AM-301 per nostril (with different spray angles)
  Other Names: Bentrio
Other: Treatment C — No treatment

SUMMARY:
Alleviation of allergic symptoms induced by house dust mites when using the medical device AM-301.

This clinical investigation explored the efficacy and safety of AM-301 when used to reduce symptoms of house dust mite sufferers. The primary objective was to compare the efficacy of AM-301 Device between treated and non-treated subjects in the treatment of perennial allergic rhinitis (PAR).

DETAILED DESCRIPTION:
This was a randomized, open-label, 3-period crossover study. The total study duration was approximately 65 days and consisted of 2 screening visits and 3 treatment visits (total 5 visits) followed by a telephone call. Patients with HDM allergy as assessed by their medical history and a positive skin prick test for Dermatophagoides pteronyssinus (der p) allergen were enrolled into the screening phase.

At least 7 days after the second screening visit, the treatment visits started. Eligible subjects were randomized to one of the six treatment sequences (ABC, BCA, CAB, ACB, BAC, CBA) at an equal ratio. The treatments were applied 10 minutes before the challenge at Visit 3, 4 and 5:

* Treatment A: One spray AM-301 (0.14 mL) per nostril,
* Treatment B: Two sprays AM-301 (0.28 mL) per nostril (at two defined spray angles in order to obtain a broader coverage of the nasal mucosa),
* Treatment C: no treatment.

The cross-over design allowed treatment C to be used as internal control. Between the three treatment visits in the chamber there was a 7±2 days wash-out period.

ELIGIBILITY:
Main Inclusion Criteria:

* Body mass index between 18.0 and 32.0 kg/m2 inclusive.
* History of perennial allergic rhinitis to house dust mite for more than 1 year.
* Positive Skin Prick Test (SPT) for Dermatophagoides pteronyssinus (der p) allergen at screening or within 12 months prior to the screening visit.

Main Exclusion Criteria:

* Any clinically relevant abnormal findings in physical examination, clinical chemistry, hematology, urinalysis, vital signs, lung function at screening visit, which, in the opinion of the investigator, may either put the subject at risk because of participation in the study or may influence the results of the study, or the subject's ability to participate in the study.
* Use of any medication considered to have an influence on the outcome of the study during the EEC session, at the discretion of the Investigator and/or designee.
* Recent nasal ulcers, mucosal erosion, nasal surgery, or nasal trauma, that might interfere with study results as determined by the Investigator and/or designee.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Couroux, MD, FRCPC, CPI, Principal Investigator — Cliantha Research
Locations (1):
- Cliantha Research, Mississauga, Canada

IPD SHARING:
Plan to Share IPD: No
Researchers may reach out to the Sponsor in order to ask for data sets.

REFERENCES:
- See also: Peer-reviewed publication of study results. PMID: 37488728 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10345461/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from November 10, 2021 (first subject first screening) to April 04, 2022 (last subject telephone call).
  Details on treatment sequences:
  Subjects that qualified for randomization, could enter the treatment period where they received a treatment before entering the chamber. This treatment could be either A - one spray of AM-301 per nostril, B - two sprays of AM-301 per nostril or C - no treatment at all. The order of the treatments was different > sequences (ABC, xxx).
Pre-assignment Details: Patients with house dust mite (HDM) allergy as assessed by their medical history and a positive skin prick test for Dermatophagoides pteronyssinus (der p) allergen were enrolled into the screening phase. 173 patients were screened and out of those, 37 patients were randomized into the prophylactic treatment phase with AM-301.
  Subjects that could not be enrolled mainly failed to show sufficient proof for HDM allergy.
Groups:
- Sequence 1: Treatment sequence for the 3 treatment visits: ABC.
- Sequence 2: Treatment sequence for the 3 treatment visits: BCA.
- Sequence 3: Treatment sequence for the 3 treatment visits: CAB.
- Sequence 4: Treatment sequence for the 3 treatment visits: ACB.
- Sequence 5: Treatment sequence for the 3 treatment visits: BAC.
- Sequence 6: Treatment sequence for the 3 treatment visits: CBA.
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 6 | 6 | 6 | 6 | 7 | 6
Completed | 5 | 6 | 5 | 6 | 5 | 6
Not Completed | 1 | 0 | 1 | 0 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol non-compliance | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Covid contact | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence 3: Treatment sequence for the 3 treatment visits:CAB.
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 6 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 7 | 6 | 37
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (8.34) | 44.8 (14.44) | 28.3 (4.84) | 40.7 (9.54) | 35.4 (10.45) | 31.7 (6.74) | 35.7 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 3 | 2 | 6 | 3 | 23
  Male | 0 | 3 | 3 | 4 | 1 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 3 | 2 | 2 | 10
  Not Hispanic or Latino | 5 | 6 | 4 | 3 | 5 | 4 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 6 | 6 | 6 | 7 | 6 | 37

OUTCOME MEASURES:

1. Primary Outcome: Overall Change From Baseline in TNSS at Visits 3, 4 and 5
Description: Total Nasal Symptom Score (TNSS) average from 20 - 180 minutes will be compared between treated and non-treated subjects. Data from all three visits are combined.
  Scale for a single symptom is from 0 - 3, 0 meaning no symptoms and 3 severe symptoms. Assessed symptoms are: nasal congestion, runny nose, nasal itching and sneezing.
  TNSS is the sum of the rating of all 4 symptoms and ranges from 0-12.
Time Frame: Day 8 to Day 22
Population: All participants received all three treatments in a different order (sequence). Therefore, data are available for each treatment for all participants. In the ITT population, all participants of the safety population with at least one TNSS assessment are included.
Measure: Mean (Standard Deviation); unit: TNSS score (0-12)
Groups:
- Treatment A: Participants received one spray of AM-301 per nostril before they entered the environmental exposure chamber (EEC).
- Treatment B: Participants received two sprays of AM-301 per nostril before they entered the environmental exposure chamber (EEC).
- Treatment C: Participants received no treatment before they entered the environmental exposure chamber (EEC).
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 36 | 36 | 34
TNSS score (0-12) | 3.9 (2.59) | 4.1 (2.93) | 5.2 (2.58)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B vs Treatment C; Treatment A + B were pooled to Treatment D for the Primary endpoint. The primary objective was to compare the efficacy of the AM-301 nasal spray (treatment D= A+B) and no treatment (C) in reducing nasal symptoms induced from HDM allergen exposure. The TNSS value from the baseline exposure (at screening exposure visit 2) was subtracted from the TNSS value of the treatment exposure to obtain change from baseline. A lower value resembles less symptoms; Test type: Superiority; p = 0.0085, ANCOVA — Treatment D (A+B) versus Treatment C

2. Secondary Outcome: Difference of Total Nasal Symptom Score (TNSS) at Individual Timepoints During House Dust Mite Challenge in the EEC (0-180 Min) Between Single and Double Application of AM-301 and no Treatment.
Description: Total Nasal Symptom Score (TNSS) average from 20 - 180 min was compared between treated and non-treated subjects.
  Scale for a single symptom is from 0 - 3, 0 meaning no symptoms and 3 severe symptoms. Assessed symptoms are: nasal congestion, runny nose, nasal itching and sneezing.
  TNSS is the sum of the rating of all 4 symptoms and ranges from 0-12.
  This descriptive endpoint was not corrected for baseline.
Time Frame: Day 8 to Day 22
Measure: Mean (Standard Deviation); unit: TNSS (0-12)
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 36 | 36 | 34
TNSS (0-12)
  Pre-chamber | 0.1 (0.35) | 0.1 (0.49) | 0.2 (0.39)
  20 min in chamber | 2.3 (2.42) | 2.4 (2.64) | 2.3 (2.25)
  40 min in chamber | 3.6 (2.71) | 3.6 (2.85) | 4.2 (3.09)
  60 min in chamber | 4.6 (2.79) | 3.6 (3.04) | 4.8 (3.42)
  80 min in chamber | 4.3 (3.05) | 4.3 (3.18) | 5.6 (2.77)
  100 min in chamber | 4.2 (2.99) | 4.7 (3.40) | 6.5 (3.08)
  120 min in chamber | 4.5 (3.06) | 4.8 (3.67) | 6.2 (3.32)
  140 min in chamber | 4.4 (3.00) | 5.1 (3.69) | 6.3 (2.96)
  160 min in chamber | 4.1 (3.33) | 4.9 (3.80) | 6.3 (3.03)
  180 min in chamber | 4.3 (3.51) | 5.1 (3.81) | 6.2 (3.32)

ADVERSE EVENTS:
Time Frame: For each participant, adverse event data were collected from day 0 to day 65 (last follow-up call).
Arm/Group | Treatment A | Treatment B | Treatment C
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/37 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/37 | 0/36
Other Adverse Events (participants affected / at risk) | 4/36 | 0/37 | 0/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=36) | Treatment B (N=37) | Treatment C (N=36)
Type I hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT05122143/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT05122143/ICF_001.pdf